CLINICAL TRIAL: NCT07327567
Title: A Randomized Clinical Trial Utilizing Crisis Response Planning in Military Personnel With Mild Traumatic Brain Injury
Brief Title: Crisis Response Planning in Military Personnel With Mild Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Hannah Tyler, Chief of Psychology, Strong Star, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001922; HT94252410714 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-12-19; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild Traumatic Brain Injury; Suicide Prevention; Suicide Risk | Patient; Suicide Risk; Suicide Risk Factor
Keywords: Clinical Response Planning; CRP; Treatment as Usual; TAU; Military personnel; suicide prevention; traumatic brain injury; TBI
MeSH Terms: conditions — Brain Concussion; Suicide Prevention; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Two-armed randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Because participants, interventionalists, and study staff cannot be blind to the behavioral therapies being delivered, only the independent evaluators will be blind to the treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Crisis Response Planning (CRP) (Experimental): One 30-60-minute session delivered individually using in-person or telehealth format by a trained behavioral health provider.
  Interventions: Behavioral: Crisis Response Planning
- Arm 2: Treatment as Usual (TAU) (No Intervention): Participants will receive the standard of care treatment as usual (TAU) from the Intrepid Spirit Center interdisciplinary treatment team that includes nurse practitioners, social workers, neurologists, and psychologists.

INTERVENTIONS:
Behavioral: Crisis Response Planning — The CRP intervention consists of a single 30-60-minute session. The CRP intervention includes a narrative assessment of the participant's most recent emotional crisis experience in order to understand and facilitate the participants understanding of their suicide mode.
  Other Names: CRP
  Arms: Arm 1: Crisis Response Planning (CRP)

SUMMARY:
The study purpose is to test the effect of Crisis Response Planning (CRP) when used as the second method of suicide prevention in military service members who are at risk for suicide due to mild traumatic brain injury (mTBI). CRP will be compared to usual treatment. The treatment will be a 30 to 60 minute session to one person at a time either in-person or using telehealth.

DETAILED DESCRIPTION:
The objective of this randomized clinical trial is to evaluate the efficacy of Crisis Response Planning as a secondary suicide prevention intervention among military service members who are at elevated risk for suicide due to their history of a mild traumatic brain injury (mTBI). CRP will be compared to a general review of available crisis resources facilitated by a therapist.

Specific Aims:

Aim 1: Determine the effectiveness of Crisis Response Planning (CRP) versus Treatment as Usual (TAU) on impulsivity and cognitive-affective states among military personnel with a diagnosis of mTBI.

Aim 2: Understand associations between impulsivity and cognitive-affective states among military personnel with a diagnosis of mTBI.

Aim 3: Determine if mTBI features (e.g., loss of consciousness duration, total number of lifetime TBIs, injury type) influence treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active duty military service members aged 18 or older.
* Diagnosis of at least one mTBI
* Ability to read, write, and speak English
* Owns and regularly uses an Apple iPhone or Android smartphone

Exclusion Criteria:

* Active psychosis as determined by clinical assessment.
* Moderate or greater cognitive impairment as indicated by evaluation by the Intrepid Spirit Center clinical team.
* Completed a Crisis Response Plan within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Beck Hopelessness Scale-5 (BHS-5) | Baseline to 3 months
  BHS is a self-report measure that assess hopelessness using a dichotomist scoring system (0 or 1).This study will use a 5-item version of the BHS developed by the Military Suicide Research Consortium. The score ranges between 0 and 5 with a higher scores indicated higher levels of hopelessness. A change in score will be reported.
Behavioral Inhibition/Activation System Scale (BIS/BAS Scale) | Baseline to 3 months
  BIS-BAS scale is a 24-item self-reporting scale for the assessment of BIS and BAS sensitivities. All items are measured on a four-point Likert scale with one indicating strong agreement and four as strong disagreements. BIS sensitivity is measured as a single factor with seven items, and the BAS sensitivity is measured as three subfactors, namely drive, reward responsiveness, and fun seeking, each measured by 4, 5, and 4 items, respectively. The scale also contains four filler items which are not scored. All the items other than two and 22 are reverse scored. A change in score will be reported.
Depressive Symptoms Index-Suicidality Subscale (DSI-SS) | Baseline to 3 months
  The DSI-SS will be used to assess current suicidal ideation. The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. Scores on each item range from 0 to 3, with higher scores reflecting greater severity of suicidal ideation. Total scores range from 0-12. A change in score will be reported.
Entrapment Scale (ES) | Baseline to 3 months
  The ES is a 16-item measure utilizes a 5-point Likert scale (0 = not at all like me; 4 = extremely like me) to evaluates both internal and external entrapment. Possible range of scores is from 0-64 with a higher score indicating greater feeling of entrapment. A change in score will be reported.
Interpersonal Needs Questionnaire-5 (INQ-5) | Baseline to 3 months
  The INQ is a self-report measure that assesses perceived burdensomeness and thwarted belongingness. This study will use a 5-item version of the INQ developed by the Military Suicide Research Consortium that showed an excellent internal consistency. Items are scored using a rating scale of 1-7 where 1=Not at all true for me to 7=Very true form me. Possible scores range from 5-35, with a higher score indicating better interpersonal relationships. A change in score will be reported.
Monetary Choice Questionnaire (MCQ) | Baseline to 3 months
  The MCQ is a 27-item, selfadministered questionnaire. For each item, the participant chooses between a smaller, immediate monetary reward and a larger, delayed monetary reward (e.g., "Would you prefer $54 today or $80 in 30 days?"). The protocol is scored by calculating where the respondent's answers place them amid reference discounting curves, with steeper curves indicating higher levels of impulsivity. A change in score will be reported.
Patient Health Questionnaire-9 (PHQ-9) | Baseline to 3 months
  The PHQ-9 is a 9-item self-report measure of the severity of depressive symptoms. Scores on the PHQ-9 have demonstrated high internal consistency and convergent validity. Items are scored from 0=Not at all to 3=Nearly every day. Total scores range from 0-27 with a higher score indicating less feeling of well-being. A change in score will be reported.
Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R_Bryan) | Baseline to 3 months
  The SITBI-R is a structured interview assessing the presence, frequency, and characteristics of self-injurious and suicidal thoughts and behaviors. The SITBI-R has high interrater reliability, strong test-retest reliability (Fox et al., 2020; Gratch et al., 2021). The SITBI-R was developed from the SITBI which also demonstrated strong psychometric properties (Nock et al., 2007). We will use the SITBI-R to measure the incidence of suicide attempts and non-suicidal self-injury.
Suicide Cognitions Scale-Revised (SCS-R) | Baseline to 3 months
  The SCS-R is a 16-item, self-report with each item scored between 0=Strongly disagree to 4=Strongly Agree. Total range of score is between 0-64 with a higher score indicating a higher level of suicidal cognition.
  measure that assesses suicide-specific thoughts and belief. The scale has demonstrated good internal consistency, convergent validity, and divergent validity (Bryan et al., 2014). The SCS-R evaluates how much an individual agrees with the suicide-related cognition. A change in score will be reported.
Temporal Experience of Pleasure Scale (TEPS) | Baseline to 3 months
  The TEPS is a 18-item self-report measure designed to assess participants' experience of positive affect using a Likert Scale from 1 (Very false for me) to 6 (Very true for me). The TEPS has strong reliability, high test-retest reliability, as well as good convergency and discriminant validity. Total possible range of score is 18-72, with a higher score indicating greater level of temporal experience of pleasure.A change in score will be reported.
Suicide - Visual Analog Scale (S-VAS). | Baseline to 3 months
  A visual analog scales with scores range from 0-100 with higher scores reflecting the higher intensity of the item being assessed (urge to die by suicide) at the moment of assessment. A change in score will be reported.
Perceived Burdensomeness - Visual Analog Scale, PB-VAS | Baseline to 3 months
  A visual analog scale with scores ranging from 0-100 with higher scores reflecting the higher intensity of the item being assessed (perceived burdensomeness) at the moment of assessment. A change in score will be reported.
Hopelessness - Visual Analog Scale (H-VAS) | Baseline to 3 months
  A visual analog scale with scores ranging from 0-100 with higher scores reflecting the higher intensity of the item being assessed (hopelessness) at the moment of assessment. A change in score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Tyler, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
As a STRONG STAR study, presentations and publications produced as a result of this work will follow the STRONG STAR Standard Operating Procedure STRONG STAR-ADM-001-5.0: Review and Approval of Publications and Presentation and the International Committee of Medical Journal Editors (ICMJE) "Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals" updated January 2024.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study completion and data are analyzed in a peer review journal and on ClinicalTrials.gov

REFERENCES:
- [Background] Bryan CJ. A Preliminary Validation Study of Two Ultra-Brief Measures of Suicide Risk: The Suicide and Perceived Burdensomeness Visual Analog Scales. Suicide Life Threat Behav. 2019 Apr;49(2):343-352. doi: 10.1111/sltb.12447. Epub 2018 Mar 7. PMID 29512832
- [Background] Di Benedetto M, Lindner H, Hare DL, Kent S. A Cardiac Depression Visual Analogue Scale for the brief and rapid assessment of depression following acute coronary syndromes. J Psychosom Res. 2005 Oct;59(4):223-9. doi: 10.1016/j.jpsychores.2005.06.070. PMID 16223625
- [Background] Huang Z, Kohler IV, Kampfen F. A Single-Item Visual Analogue Scale (VAS) Measure for Assessing Depression Among College Students. Community Ment Health J. 2020 Feb;56(2):355-367. doi: 10.1007/s10597-019-00469-7. Epub 2019 Sep 17. PMID 31531784
- [Background] Kertzman S, Aladjem Z, Milo R, Ben-Nahum Z, Birger M, Grinspan H, Weizman A, Kotler M. The utility of the Visual Analogue Scale for the assessment of depressive mood in cognitively impaired patients. Int J Geriatr Psychiatry. 2004 Aug;19(8):789-96. doi: 10.1002/gps.1141. PMID 15290703
- [Background] Bryan CJ, David Rudd M, Wertenberger E, Etienne N, Ray-Sannerud BN, Morrow CE, Peterson AL, Young-McCaughon S. Improving the detection and prediction of suicidal behavior among military personnel by measuring suicidal beliefs: an evaluation of the Suicide Cognitions Scale. J Affect Disord. 2014 Apr;159:15-22. doi: 10.1016/j.jad.2014.02.021. Epub 2014 Feb 19. PMID 24679384
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Gratch I, Fernandes SN, Bell KA, Pollak OH, Fox KR, Tezanos K, Ebo T, Cha CB. Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R): Reliability, Validity, and Inter-Informant Agreement in an Adolescent Sample. J Clin Child Adolesc Psychol. 2022 Jul-Aug;51(4):484-494. doi: 10.1080/15374416.2021.1901229. Epub 2021 Apr 13. PMID 33847199
- [Background] Fox KR, Harris JA, Wang SB, Millner AJ, Deming CA, Nock MK. Self-Injurious Thoughts and Behaviors Interview-Revised: Development, reliability, and validity. Psychol Assess. 2020 Jul;32(7):677-689. doi: 10.1037/pas0000819. Epub 2020 Apr 23. PMID 32324021